CLINICAL TRIAL: NCT03486262
Title: Lung Cancer and Idiopathic Pulmonary Fibrosis : Pathological and Molecular Characterization
Acronym: K-FPI
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI16034
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-02

CONDITIONS: Lung Cancer and Idiopathic Pulmonary Fibrosis
Keywords: Lung cancer; Idiopathic pulmonary fibrosis
MeSH Terms: conditions — Lung Neoplasms; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Formalin fixed paraffin embedded lung samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung carcinoma on IPF: Lung carcinoma on IPF

SUMMARY:
Retrospective inclusion of lung cancers developed in a context of idiopathic pulmonary fibrosis, diagnosed and / or treated in participating centers. The cases are recovered retrospectively from the records of the pulmonology and pathology departments of our various partners.

DETAILED DESCRIPTION:
Primary objective:

Characterize altered molecular pathways in lung cancer in patients with IPF versus lung cancer in non-IPF patients.

Secondary objectives:

Identify specific therapeutic targets Describe a cohort of lung cancers on IPF (clinical / radiological and pathological data) To study the relationship between neoplastic / preneoplastic lesions and pulmonary parenchyma reshaped by fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Lung carcinoma
* Idiopathic pulmonary fibrosis

Exclusion Criteria:

- No tumor sample available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective inclusion of lung cancers developed in a context of idiopathic pulmonary fibrosis, diagnosed and / or treated in participating centers. The cases are recovered retrospectively from the records of the pulmonology and pathology departments of our various partners.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Molecular profile of IPF-associated lung carcinomas | 1 month / 8 samples
  Next generation sequencing of carcinomas with Ion S5 XL sequencer and Oncomine™ Comprehensive Panel

SECONDARY OUTCOMES:
Pathological characterization of lung carcinomas | 1 month / 8 samples
  Histological classification of carcinomas and immunohistochemistry with lineage markers

CONTACTS AND LOCATIONS:
Overall Officials: Auréie CAZES, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital BICHAT-CLAUDE BERNARD, Paris, France